CLINICAL TRIAL: NCT02004431
Title: A Case-control Study of Peri-operative Psychological State and Acute and Chronic Post-operative Pain
Brief Title: Peri-operative Psychology and Post-operative Pain Study
Acronym: 4P
Status: Completed | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 13/P/159; 137267 (Other: IRAS)
Record Dates: First submitted 2013-11-11; First posted 2013-12-09 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2014-09

CONDITIONS: Surgery; Pain; Anxiety; Depression
Keywords: Chronic post surgical pain; Orthopaedic; Anxiety; depression
MeSH Terms: conditions — Pain; Anxiety Disorders; Depression; Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pain (experimental): The cases are patients with significant pain on day one after surgery
- No pain (control): The controls are sex, age and operation matched individuals without pain.

SUMMARY:
The experience of pain is common among hospital inpatients. Orthopaedic surgery often results in significant pain, which may last for some time. About one in eight people will experience long-term or chronic pain after surgery, which can impact on quality of life and mood. Some risk factors are known for chronic post surgical pain (CPSP) and these include patient factors, surgical factors and anaesthetic factors. We know that mood problems (anxiety and depression) increase the risk of CPSP. What is not known is how short term changes in mood are related to the experience of pain after surgery and how this impacts on CPSP. This study is designed to investigate the relationship between both short and long-term mood problems and short and long-term pain and quality of life after orthopaedic surgery. The study will provide valuable information to allow us to design a psychological intervention, which might reduce the risk of short-term post surgical pain and CPSP.

This study also aims to measure a number of other variables, which may be related to CPSP including medication use, other medically unexplained symptoms and catastrophic thinking in response to pain.

All patients having planned orthopaedic surgery will be asked to enter the trial. Those consenting to involvement will complete a questionnaire assessing the variables described above. They will be divided into two groups depending on whether they have significant pain on the day after their surgery. As the primary aim of the study, the rates of significant anxiety or depression will then be compared between these two groups.

Secondary outcomes will be assessed by a questionnaire sent to the patients at 6 months after their surgery. Descriptive statistics will be produced for all the variables and use to model a future study, which would assess the effect of a psychological intervention on acute and chronic post surgical pain.

Our hypothesis is that patients are more likely to experience acute anxiety and depression or display catastrophic thinking if they suffer significant post-surgical pain. The study is powered to reliably detect a three-fold difference in the prevalence of psychopathology between patients with and without acute pain on day 1 after elective orthopaedic surgery.

DETAILED DESCRIPTION:
This is a prospective case-control observational study. The primary aim is to determine whether patients with poor pain control on day 1 following surgery have higher levels of anxiety / depression or catastrophising than those without acute pain. The cases are patients with significant pain on day one after surgery and the controls are sex, age and operation matched individuals without pain.

Several other variables are measured which may provide information for the design of future studies. The presence of pain or psychopathology prior to surgery will be recorded, as this is likely to impact on these variables in the post-operative period. Analgesic use pre and post surgery is also of interest as a surrogate measure of pain severity.

In addition to day one data, pain severity will also be recorded on day 2 and 3 post-operatively. This is of interest as although most patients will be expected to demonstrate reducing pain severity with time, a proportion will not improve and a small number will experience increasing pain with time. This adverse "pain trajectory" might be associated with an increased incidence of CPSP 28.

Long-term outcomes such as pain and quality of life at 6 months post-discharge will also be assessed by postal questionnaire.

The eventual aim of this series of studies is to assess the interaction between acute psychological problems and post-surgical pain and the impact that this has on longer-term outcomes such as CPSP, mood and quality of life. Short-term pre- and post-operative psychological interventions will then be developed to modify the impact of psychological factors on long-term surgical outcomes. Further studies will assess the efficacy of these interventions. Pre-study audit will be carried out to confirm the feasibility of matching.

ELIGIBILITY:
Inclusion Criteria:

* All inpatients on Sharp, Shaugh or Stannon ward following elective orthopaedic surgery carried out on Monday to Thursday each week.

Exclusion Criteria:

* Patient refusal, Age <18, Emergency / trauma surgery, Day case surgery, unable to read or understand written instructions, No contact address, Not registered with a General Practitioner (GP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of all patients following elective orthopaedic surgery with a planned inpatient stay of at least 24 hours
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Is acute pain following orthopaedic surgery is associated with the onset of anxiety as measured using the Generalised Anxiety Disorder Questionnaire (GAD-7) | 24 hours
  This is a prospective case-control observational study. The primary aim is to determine whether patients with poor pain control on day 1 following surgery have higher levels of anxiety than those without acute pain. The cases are patients with significant pain on day one after surgery and the controls are sex, age and operation matched individuals without pain.
Is acute pain following orthopaedic surgery is associated with the onset of depression as measured using the Patient Health Questionnaire (PHQ-9). | 24 hours
  This is a prospective case-control observational study. The primary aim is to determine whether patients with poor pain control on day 1 following surgery have higher levels of depression than those without acute pain. The cases are patients with significant pain on day one after surgery and the controls are sex, age and operation matched individuals without pain.
Is acute pain following orthopaedic surgery is associated with the onset of abnormal coping strategies as measured using the Pain Catastrophising Scale (PCS). | 24 hours
  This is a prospective case-control observational study. The primary aim is to determine whether patients with poor pain control on day 1 following surgery have higher levels of catastrophising than those without acute pain. The cases are patients with significant pain on day one after surgery and the controls are sex, age and operation matched individuals without pain.

SECONDARY OUTCOMES:
Acute pain (NRS) will be measured on day 1 after surgery. | 24 hours
  Correlation between acute variables (pain, anxiety, depression and catastrophising) will be sought with length of hospital stay and the presence of chronic post surgical pain at 6 months
Acute post operative pain (NRS) at 6 months | 6 months
  Correlation between acute variables (pain, anxiety, depression and catastrophising) will be sought with length of hospital stay and the presence of chronic post surgical pain at 6 months.
  Correlation will be sought between pain immediately after surgery and chronic post surgical pain 6 months later.
  Acute pain, anxiety & depression will be measured in day 1 post operatively and correlated with quality of life at 6 months (EQ5D).
Pre operative strong opioid use (binary variable) | 24 hours
  To test any association between pre-operative strong opioid use and acute or chronic post surgical pain and continued opioid use at 6 months.
Total opioid intake before surgery | 24 hours
  Correlation between acute anxiety, depression or catastrophising and total opioid intake before and 1 day & 6 months after surgery
Somatic symptoms questionnaire (bespoke questionnaire) | 24 hours
  This questionnaire records other somatic symptoms patients may experience and the total score will be used to determine any correlation with acute psychopathology, pain and outcomes following surgery as described above.
Perception of care questionnaire (bespoke questionnaire) | 24 hours
  This questionnaire contains details of the inpatient experience and we will investigate whether patient perceptions of care correlate with psychopathology, pain and outcomes following surgery
Anxiety (GAD7) will be measured on day 1 after surgery. | 24 hours
  Correlation between acute variables (pain, anxiety, depression and catastrophising) will be sought with length of hospital stay and the presence of chronic post surgical pain at 6 months.
  PHQ9 & GAD 7 scores on day 1 after surgery and at 6 months. Presence of treated anxiety or depression before surgery (binary score). The frequency of significant anxiety or depression will be compared before and after surgery
Depression (PHQ9) will be measured on day 1 after surgery. | 24 hours
  Correlation between acute variables (pain, anxiety, depression and catastrophising) will be sought with length of hospital stay and the presence of chronic post surgical pain at 6 months.
  PHQ9 & GAD 7 scores on day 1 after surgery and at 6 months. Presence of treated anxiety or depression before surgery (binary score). The frequency of significant anxiety or depression will be compared before and after surgery
Catastrophising (PCS - pain catastrophising scale) will be measured on day 1 | 24 hours
  Correlation between acute variables (pain, anxiety, depression and catastrophising) will be sought with length of hospital stay and the presence of chronic post surgical pain at 6 months
Acute anxiety (GAD7) | 6 months
  Acute pain, anxiety & depression will be measured in day 1 post operatively and correlated with quality of life at 6 months (EQ5D)
Depression (PHQ9) | 6 months
  Acute pain, anxiety & depression will be measured in day 1 post operatively and correlated with quality of life at 6 months (EQ5D)
Quality of life (EQ5D) | 6 months
  Acute pain, anxiety & depression will be measured in day 1 post operatively and correlated with quality of life at 6 months (EQ5D)
Opioid use at 6 months (binary variable) | 6 months
  To test any association between pre-operative strong opioid use and acute or chronic post surgical pain and continued opioid use at 6 months.
Total opioid intake on day 1 post surgery | 24 hours
  Correlation between acute anxiety, depression or catastrophising and total opioid intake before and 1 day & 6 months after surgery
Length of hospital stay (days) | Days
  Correlation between acute variables (pain, anxiety, depression and catastrophising) will be sought with length of hospital stay and the presence of chronic post surgical pain at 6 months
Catastrophising (PCS - pain catastrophising scale) | 6 months
  Acute pain, anxiety & depression will be measured in day 1 post operatively and correlated with quality of life at 6 months (EQ5D)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rockett, MB ChB, PhD, Principal Investigator — University Hospital Plymouth NHS Trust
Locations (1):
- Plymouth Hospitals NHS Trust, Plymouth, Devon, United Kingdom